CLINICAL TRIAL: NCT05063253
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy of TG103 Injection in Overweight/Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of TG103 Injection in Overweight/Obese Subjects With Type 2 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSA1803-CSP-006
Record Dates: First submitted 2021-09-14; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TG103, 15 mg (Experimental): TG103 (15 mg) will be administered via subcutaneous injection once weekly.
  Interventions: Drug: TG103
- TG103, 22.5 mg (Experimental): TG103 (22.5 mg) will be administered via subcutaneous injection once weekly.
  Interventions: Drug: TG103
- TG103, 30 mg (Experimental): TG103 (30 mg) will be administered via subcutaneous injection once weekly.
  Interventions: Drug: TG103
- Placebo (Placebo Comparator): Placebo will be administered via subcutaneous injection once weekly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TG103 — TG103 injection, SC, once weekly
  Other Names: Administered SC
  Arms: TG103, 15 mg; TG103, 22.5 mg; TG103, 30 mg
Drug: Placebo — Placebo, SC, once weekly
  Other Names: Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy, safety, PK and PD characteristics of different doses of TG103 injection in overweight/obese subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy of TG103 injection in subjects with type 2 diabetes mellitus combined with overweight/obesity. The study will consist of 3 periods: an approximately 4-week screening period, a 20-week treatment period, and a 3-week safety follow-up period. Eligible subjects will be randomized in a 1:1:1:1 ratio into four paralleled dose groups (15 mg, 22.5 mg ,30 mg and placebo) with 52 subjects in each group. Within each group, subjects will receive TG103 injection or placebo subcutaneously (SC) once a week (QW) over a period of 20 weeks. Each group will be started at a low dose of 7.5 mg and gradually up-titrated at weekly intervals until the target dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have diagnosed with type 2 diabetes according to the Guidelines for prevention and treatment of type 2 diabetes in China (2020 Edition);
2. Aged 18 to 75 years (inclusive), no gender limitation;
3. Body mass index (BMI) ≥ 24.0 kg/m^2 with stable body weight (less than 5% self-reported change within 3 months);
4. Subjects diagnosed with type 2 diabetes ≤ 3 years, and not on medication or with a history of regular medication for no more than 1 week within the 3 months prior to screening (subjects with a history of medication only include those with a history of single-agent oral medication and a history of short-term intensive insulin therapy (≤ 2 weeks)); 5.7.5% ≤ HbA1c ≤ 10.0%;

6.Subjects of childbearing potential must use reliable methods of contraception from the date of signing an informed consent to at least 3 months after the last dose; 7. The subject fully understand the trial and possible adverse reactions, has the ability to communicate properly with the investigator and comply with the research protocol; 8.Voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Fasting plasma glucose ≥ 13.9 mmol/L at screening or a history of severe hypoglycemia (Serious event requiring help from others with changes in consciousness and/or body) within 6 months prior to screening;
2. Systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg during screening;
3. Have one or more positive tests in anti-human immunodeficiency virus antibody or anti-treponema pallidum-specific antibody;
4. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≥2.5x upper limit of normal (ULN), or Total bilirubin (TBiL)≥1.5x ULN, or triglyceride > 5.7 mmol/L or eGFR < 60 mL/(min*1.73 m^2) during the screening period;
5. Subjects with hematological diseases (e.g., aplastic anemia, myelodysplastic syndrome) or any disease causing hemolysis or erythrocyte instability (e.g., malaria), or hemoglobin<100 g/L;
6. Hypercortisolism, polycystic ovary syndrome, abnormal thyroid function (those requiring medication or who have not reached a stable dose of treatment in 3 months prior to screening), etc. or other diseases that may affect blood glucose metabolism;
7. Have a personal or family history of medullary thyroid carcinoma (MTC) or type 2 multiple endocrine neoplasia, or other genetic diseases that are susceptible to medullary cancer, or calcitonin ≥ 50 ng/L(pg/mL);
8. Acute complications of diabetes (including diabetic ketoacidosis, hyperosmolar nonketotic diabetic coma, lactic acidosis) occurred once or more within 3 months or twice or more within 6 months before screening;
9. Proliferative diabetic retinopathy, foot ulcers/gangrene, and manifestations of peripheral neuropathy with obvious symptoms (e.g., gastroparesis, urinary retention, intestinal obstruction, urinary incontinence, and painful peripheral neuropathy);
10. Subjects with degree II or III atrioventricular block in 12-lead ECG (except for subjects who use the pacemaker), long QT syndrome or prolonged QTc interval (QTcF: >450 ms for males, >470 ms for females), or signs of clinically significant localised ischemic heart disease during the screening period; or those with other heart diseases that are judged by the investigator to be unsuitable for entry into the study;
11. Any of the following cardiovascular and cerebrovascular events within half a year before screening: unstable angina pectoris requiring hospitalization, myocardial infarction, coronary artery bypass grafting, percutaneous coronary intervention (diagnostic angiography is allowed), moderate to severe congestive heart failure (NYHA grade III or IV), atrial or ventricular arrhythmia requiring hospitalization (such as atrial fibrillation and ventricular tachycardia), pacemaker or defibrillator implantation, transient ischemic attack or cerebrovascular accident (e.g. stroke), or those with coronary artery bypass grafting or revascularization planned during the study period;
12. Have chronic or acute pancreatitis ( or have a history of recurrent acute pancreatitis), or serum amylase and/or lipase ≥ 3x ULN (If lipase cannot be detected in some centers, it is acceptable to judge only based on amylase),or severe gastrointestinal disease, such as confirmed reflux esophagitis or gallbladder disease, or any disease impacting gastric emptying (such as gastric bypass surgery, pyloric stenosis, except for appendectomy) or gastrointestinal diseases that may be aggravated by GLP-1 analogues; for subjects with a history of gallbladder stones (gallstone removal or lithotripsy) and/or cholecystectomy, access to the study will be determined by investigator after assessing the risk if there are no further sequelae;
13. History of severe respiratory tract, blood system, central nervous system diseases (e.g., epilepsy, etc.), or history of malignant tumor (except for basal cell carcinoma or carcinoma in situ that has been clinically cured), mental diseases (e.g., depression, anxiety, etc.), or history of other diseases that may endanger the safety of the subjects and are considered unsuitable for this study in the investigator's opinion;
14. Subjects who have undergone major surgery within 3 months before screening, or have ongoing severe or acute infection within 4 weeks before screening, or whose white blood cell count exceeds 10% of the upper limit of normal during the screening period;
15. Use of drugs that can affect glucose metabolism or directly reduce gastrointestinal motility within the 3 months prior to screening or expected during the course of the study, including the cumulative use of systemic glucocorticoids (topical, intraocular and inhaled preparations), immunosuppressants and cytotoxic drugs for more than 7 days; Large doses of thiazide diuretics (hydrochlorothiazide>100 mg/d, chlorothiazide> 2 g/d, indapamide> 5 mg/d, chlorthalidone> 100 mg/d), anticholinergics, antispasmodics, etc. for more than 7 consecutive days;
16. Have taken prescription or over-the-counter medications for weight loss (e.g., orlistat, sibutramine, rimonabant, phenylpropanolamine, or chlorphenimiindole, etc) within 3 months prior to screening; or have undergone surgery that can cause weight instability;
17. Drugs that may cause significant weight gain have been used or are being used within 3 months before screening, including tricyclic antidepressants, atypical antipsychotics and mood stabilizers (e.g., midazolam, amitriptyline, mirtazapine, paroxetine, phenyl valproic acid and its derivatives and lithium), etc;
18. Have a serious history of drug or food allergy, or may be allergic to the investigational product according to the judgment of the investigator;
19. Lost more than 400 mL of blood due to blood donation or other reasons within 3 months before the screening period;
20. Average alcohol intake more than 21 units of alcohol (male)/14 units of alcohol (female) per week within the 3 months prior to screening;
21. Regular consumption of caffeine more than 600 mg per day within the 3 months prior to screening;
22. Smoke more than 20 cigarettes per day within 3 months prior to screening;
23. Have skin abnormalities or dermatitis within a radius of 2 cm of the administration site;
24. Participation in other drug studies within 3 months prior to screening and the last received test drug less than 3 months prior to screening; or subjects out of the group due to adverse events in the previous study; or attempted to participate in other drug trials during the study;
25. Pregnant (blood pregnancy test positive in screening period) or lactating female;
26. Vaccinated within 28 days before screening or planned to be vaccinated during the study;
27. Not suitable for this study in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Changes in glycosylated hemoglobin (HbA1c) from baseline to week 20 | Baseline through Day 141 (the end of the 20-week treatment)

SECONDARY OUTCOMES:
Change in body weight from baseline to week 20 | Baseline through Day155 (the end of the follow-up)
Change in body mass index (BMI) from baseline to week 20 | Baseline through Day155 (the end of the follow-up)
Change in waist circumference from baseline to week 20 | Baseline through Day155 (the end of the follow-up)
Change in waist-hip ratio from baseline to week 20 | Baseline through Day155 (the end of the follow-up)
Change in blood pressure(systolic and diastolic blood pressure) from baseline to week 20 | Baseline through Day155 (the end of the follow-up)
Change in blood lipid from baseline to week 20 | Baseline through Day155 (the end of the follow-up)
Proportion of subjects with a baseline weight loss of more than 5% | Baseline through Day155 (the end of the follow-up)
Incidence of adverse events | Baseline through Day155 (the end of the follow-up)
Minimum steady-state plasma drug concentration during a dosage interval (Cmin, SS) | Day1, 29, 57, 85 and 113
Change in fasting blood glucose from baseline to week 20 | Baseline through Day 141 (the end of the 20-week treatment)
Change in 2-hour postprandial blood glucose from baseline to week 20 | Baseline through Day 141 (the end of the 20-week treatment)
The occurrence of TG103 anti-drug antibodies (ADA) and neutralizing antibody (Nab). | Day1, 29, 57, 85, 113 and 155

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School

IPD SHARING:
Plan to Share IPD: No